CLINICAL TRIAL: NCT06557226
Title: Oral (Hypo-)Function, General Function and Nutritional Status in Elderly Hospitalized Patients
Acronym: Ohyp
Status: Completed | Type: Observational
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Frauke Müller, Professor, University of Geneva, Switzerland
Other Study IDs: 2019-01338
Record Dates: First submitted 2024-07-01; First posted 2024-08-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Oral Health; Oral Health Related Quality of Life; Nutrition Disorders in Old Age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patient with oral hypofunction with 3 impaired oral functional parameters: patient's will receive an oral examination comprising the evaluation of 7 parameters: the oral hygiene, the oral dryness, the occlusal force, the tongue-lip motor function, the tongue pressure, the chewing function and the swallowing function. Oral hypofunction is defined as a state when 3 or more signs were present.
  Interventions: Other: oral and nutritional examination

INTERVENTIONS:
Other: oral and nutritional examination — Participants will receive a comprehensive oral examination, nutritional examination and will fill an oral health related quality of life questionnaire.

SUMMARY:
The goal of this observational study is to learn about the effects of a reduced oral function on the nutritional status of non-acute hospitalized elders and on their oral health quality of life.

DETAILED DESCRIPTION:
Malnutrition is highly prevalent among the elderly, many authors reported on the relationship between oral health and nutrition. However the the relationship between the dental state and the nutritional status was always limited to anatomical criteria such as number of teeth and the presence of prosthetic reconstructions.

The oral function is classified into 4 stages healthy state, oral frailty, oral hypofunction and oral dysfunction. The classification into the different stages result from an examination of 7 parameters: the oral hygiene, the oral dryness, the occlusal force, the tongue-lip motor function, the tongue pressure, the chewing function and the swallowing function.

This study aims to correlate the oral function with the nutritional status of non-acute hospitalized elders. And to further investigate the correlation between the different parameters defining the oral function and the oral health related quality of life (OHRQoL) as measured by theGeneral Oral Health Assessment Index.

A total 60 participants will be recruited in the University Hospital of Geneva, Loëx rehabilitation center. The investigators will see the patient for 2 visits after informed consent. The first visit will be 45 minutes long and will include a dental examination and an examination of the oral hygiene, the oral dryness, the tongue lip motor function, the tongue pressure, the occlusal force and the swallowing function. Diagnosis for nutrition according to the Glim criteria will be done. Furthermore, the participants will be asked to fill an oral health quality of life questionnaire comprising 12 questions.

Oral hypo function will be defined as a state when 3 or more signs were present from the 7 parameters examined.

Linear multiple regression analysis is used to examine the relationship between the nutritional status and oral function. Spearman's rank correlation coefficient will be used to correlate the oral function score and oral health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* • Aged 70 years or over

  * Hospitalized in Geneva University Hospitals, in rehabilitation or in long term care (Loëx)
  * Able to follow simple instructions and perform the tests
  * Understand French and complete or answer the questionnaire
  * Give written informed consent
  * Consent can be obtained from their next of kin or legal representative if necessary
  * Have been admitted into the hospital no longer 15 days before inclusion

Exclusion Criteria:

* Patients with tube/intravenous feeding
* Poorly-controlled diabetes (Liu et al., 2015)
* Patients with gastro-intestinal diseases or symptoms (nausea, vomiting, diarrhea, constipation) affecting oral intake
* If the patient is taking an antimicrobial treatment at this time.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will enroll 60 patients aged 70 years or more and admitted to the Geneva University Hospitals (HUG) at Loëx Hospital. Patients will be approached consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Malnutrition status as classified by the Global Leadership Initiative on Malnutrition (GLIM) | baseline
  The GLIM considers both (a) phenotypic (>5% weight loss within the previous 6 months or >10% weight loss in more than 6 months, BMI < 22 kg/m2 if age >70 years, FFMI <17 kg/m2 in men and <15 kg/m2 in women) and (b) aetiologic criteria (reduced food intake and level of inflammation with CRP >10 mg/L). Participants were classified as malnourished when at least 1 phenotypic criterion and 1 aetiologic criterion were met. The severity of the malnutrition is based on the phenotypic criteria in a stage 1 "moderate malnutrition" and stage 2 "severe malnutrition." The participants were classified on a score scale from 0- 2 with o being normal, 1 for the moderate malnutrition and 2 for the severe malnutrition.
Number of impaired oral functions | baseline
  The Japanese society of gerodontology in 2016 published a position paper aiming to standardize the examination of oral disorders related to age and to suggest management strategies. They created a conceptual diagram divided into 4 stages: healthy state, oral frailty, oral hypofunction and oral dysfunction. The classification into the different stages result from an examination of 7 parameters: the oral hygiene, the oral dryness, the occlusal force, the tongue-lip motor function, the tongue pressure, the chewing function and the swallowing function. Oral hypofunction is defined as a state when 3 or more signs were present.

SECONDARY OUTCOMES:
Oral health related quality of life | baseline
  General oral health assessment index (GOHAI) is a self-reported measure designed to assess the impact on daily life of oral health problems of older individuals. The 12 item GOHAI evaluates three dimensions of oral health related quality of life study (OHRQOL).
  The GOHAI score is determined by summing the final score of each of the 12 items ranges from 0 to 60 with higher scores indicating better oral health.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Graf, Pr., Study Director — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - University clinics of dental medicine, Geneva, Canton of Geneva
  - Geneva University Hospital, Geneva, Canton of Geneva

IPD SHARING:
Plan to Share IPD: Undecided